CLINICAL TRIAL: NCT02222298
Title: Video Assisted Ablation of Pilonidal Sinus Versus Convention Off-midline Bas Com Cleft Lift Procedure
Brief Title: Video Assisted Ablation of Pilonidal Sinus Versus Conventional Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Francesco Milone, Professor of Surgery, Federico II University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: framar
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Sacrococcygeal Pilonidal Sinus

ARMS (2):
- VAAPS group (Experimental): patients undergoing video assisted ablation of pilonidal sinus
  Interventions: Procedure: Video assisted ablation of pilonidal sinus
- conventional treatment group (Active Comparator): patients undergoing conventional off-midline Bascom cleft lift procedure
  Interventions: Procedure: Bascom Cleft lift procedure

INTERVENTIONS:
Procedure: Video assisted ablation of pilonidal sinus — A 5-phases' technique. The 1st phase is to insert the endoscope through the external opening (orifice). In the patients that had more than one opening the lower pit is used for access. The 2nd phase is to identify the sinus cavity and its lateral tracks. The endoscope is advanced along the pathway using slow movements, left/right and up/down. These manoeuvres and the saline solution, used as distension medium, allow the sinus cavity to accommodate the endoscope. Additionally mechanical adhesiolysis with the forceps grasping could be useful. The 3rd phase is to identify the presence of hair and its removal. The 4th phase phase is to obtain complete ablation of sinus cavity. The sinus cavity and its lateral tracks are destroyed with the electrode under continuous direct vision. The 5th phase is to obtain the accurate cleaning of sinus cavity. The saline solution flow allows the elimination of any necrotic material. A Volkmann spoon could be useful to complete the cleaning.
  Arms: VAAPS group
Procedure: Bascom Cleft lift procedure
  Arms: conventional treatment group

SUMMARY:
Video assisted ablation of pilonidal sinus (VAAPS) is a new endoscopic minimally invasive treatment. In an attempt to validate the effectiveness of the VAAPS, the investigators have designed a comparative study between the conventional and the minimally invasive treatment. Two surgical procedures were evaluated: VAAPS (Experimental group) and conventional excision with a Bascom out-midline closure (Control group).

ELIGIBILITY:
Inclusion Criteria:

* Chronic sacrococcygeal pilonidal sinus

Exclusion Criteria:

* Absence of consent to the study
* Acute abscess

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Infection | at 30 days after surgery
  Wound infection was defined as redness and/or oedema of the skin and/or discharge.

SECONDARY OUTCOMES:
recurrence | at 1 year after surgery
  recurrence was defined when symptoms of the disease recurred after an interval following complete wound healing.
return at work | up to 30 days after surgery
Pain | up to 30 days after surgery
  A vas-score scale (0-10) will be used
satisfaction | up to six months after surgery
  a Vas-score scale (0-10) and a SF_36 model will be used

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples "Federico II", Naples, Italy, Italy